CLINICAL TRIAL: NCT02308397
Title: Bakery Products for Non-Coeliac Gluten Sensitive Consumers
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Aberdeen (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Other
Other Study IDs: Rowett 904
Record Dates: First submitted 2014-11-13; First posted 2014-12-04 (Estimated); Last update posted 2017-10-27 (Actual); Status verified 2017-10

CONDITIONS: Non Coeliac Gluten Sensitivity
Keywords: non coeliac gluten sensitivity; gluten; bread
MeSH Terms: interventions — Bread

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Group 1 (Experimental): Begins with Normal gluten containing bread
  Interventions: Other: Normal gluten containing bread
- Group 2 (Experimental): Begins with Bread with reduced gliadins content
  Interventions: Other: Bread with reduced gliadins content
- Group 3 (Experimental): Begins with Bread with reduced ATIs content
  Interventions: Other: Bread with reduced ATIs content
- Group 4 (Experimental): Begins with Bread with reduced overall protein content
  Interventions: Other: Bread with reduced overall protein content

INTERVENTIONS:
Other: Normal gluten containing bread — Group 1 will begin with Normal gluten containing bread(A) and then move to bread B,C and D
  Arms: Group 1
Other: Bread with reduced gliadins content — Group 2 will begin with Bread with reduced gliadins content (B) and then move to bread A, C and D
  Arms: Group 2
Other: Bread with reduced ATIs content — Group 3 will begin with Bread with reduced ATIs content (C) and then move to bread A, B and D
  Arms: Group 3
Other: Bread with reduced overall protein content — Group 4 will begin with Bread with reduced overall protein content (D) d then move to bread A, B and C
  Arms: Group 4

SUMMARY:
The aim of the study is to produce a tolerable alternative to normal wheat bread which would be suitable for subjects with self-reported non-coeliac gluten sensitivity (NCGS). The bread would be made from wheat so, in contrast to gluten-free bread, would be more comparable to standard bread. To make this bread, the investigators will use advanced enzyme technology and/or novel formulations to target the digestion or removal of wheat proteins, which might be involved in the etiology of non-coeliac gluten sensitivity, preferentially over other those that are more useful for baking quality. The investigators will determine palatability and tolerance of this new product in a human cross-over, randomised, blind and placebo-controlled intervention study.

It has been estimated 6-10% of the population are sensitive to gluten who do not have coeliac disease (CD). Three breads will be produced and tested in this study against a suitable reference based on standard wheat flour and baking process

DETAILED DESCRIPTION:
Prior to the study each volunteer will undergo screening procedure (Health Screening Questionnaire) for compliance with the inclusion/exclusion criteria. The volunteers who meet those criteria will be invited to sign an informed consent. Following this the volunteers will be asked to complete:

* Gluten Sensitivity Questionnaire
* SF-36 Quality of Life Questionnaire
* Beacke Physical Activity Questionnaire
* DASS 21 Questionnaire

It is anticipated that NCGS volunteers are following a low gluten or gluten-free life style. Evaluation of their dietary compliance with gluten-free diet will be done through using numerical scores (Biagi at al.,2009) - a system based on strategies that the subjects use to avoid eating gluten.

Gastrointestinal symptoms will be assessed by the participant completing daily diary cards via a 100-mm VAS to score the presence and severity of overall abdominal symptoms, abdominal pain, bloating, wind, satisfaction with stool consistency, tiredness, and nausea.

Severity of fatigue will be evaluated by the Daily-Fatigue Impact Scale (D-FIS), a questionnaire containing 8 items that evaluates the impact of fatigue on cognition, physical functioning, and daily activities.

After one week of a baseline period, the subjects will be assigned to one week of dietary intervention (bread A, B, C or D), followed by 14-day wash-out period before crossing over to the next bread. All volunteers will be randomised to all four groups/cross over intervention.

Treatment:

* Bread A - normal (gluten-containing) reference bread
* Bread B - bread with reduced gliadin content
* Bread C - bread with reduced ATIs
* Bread D - bread with reduced overall protein content

Each treatment bread will be consumed for one week (3 slices per day), followed by washout period of at least 2 weeks or until symptoms induced during the previous dietary challenge resolved. Volunteers unable to continue a treatment due to intolerable symptoms will be permitted to cease the study food of that particular arm but can continue if they wish with the study.

Bread will be provided to volunteers at the beginning of each treatment week. Compliance will be determined with questioning at time of review and counting the slices of bread left at the end of the treatment week.

Pilot study

For volunteers only recruited from the Aberdeen and the Aberdeenshire area as part of a pilot study we will also ask volunteers to make a single visit (at the beginning of the study) to the RINH. At this visit a fasting blood sample will be taken, the blood pressure will be checked and anthropometric measurements will be made.

Blood test:

* IgA anti-tissue transglutaminase antibody and total IgA level.
* IgA endomysial antibody
* IgG deamidated gliadin peptide antibodies (DGP-AGA)
* Immunoglobulin IgG/IgA antigliadin antibodies (AGA)
* Flow cytometric basophil activation test
* Gliadin-specific T cells in the peripheral blood
* Full blood count
* Lipid profile
* Vit B12 and folic acid status

ELIGIBILITY:
Inclusion Criteria:

* male or female, aged 18-70, who believe they experience non-coeliac gluten sensitivity

Exclusion Criteria:

* Medical exclusion criteria

  * Coeliac Disease
  * Wheat allergy
  * Dermatitis Herpetiformis
  * Gastrointestinal disorders: Small Intestinal Bowel Overgrowth (SIBO), Crohn's disease , Ulcerative Colitis, Inflammatory Bowel Disease (IBD)
  * History of gastrointestinal surgery/procedure over the last 3 years
  * Kidney disease
  * Hepatic disease
  * Active cancer
  * Severe cardiovascular disease
  * Addiction to any substances
  * Breastfeeding/ Pregnancy

Volunteers with poorly controlled psychiatric disease or those unable to give written informed consent will also be excluded.

Medication exclusion criteria

* Medications for treatment of heartburn, dyspepsia, indigestion, bloating etc. e.g. gastrokinetics or prokinetics, antacids, laxatives
* Digestive enzymes

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2014-11; Primary Completion 2018-03 (Estimated); Study Completion 2018-03 (Estimated)

PRIMARY OUTCOMES:
Change in the presence and severity of overall and individual gastrointestinal symptoms (daily diary cards via a 100-mm VAS to score) | These will be assessed daily during baseline week (0), treatment week (1, 4, 7 and 10) and washout week (3, 6 and 9)
  Gastrointestinal symptoms will be assessed by the participant completing daily diary cards via a 100-mm VAS to score the presence and severity of abdominal pain, bloating, wind and nausea.

SECONDARY OUTCOMES:
Change in the presence and severity of daily fatigue (Daily-Fatigue Impact Scale (D-FIS) | Fatigue will be assessed daily during baseline week (0), treatment week (1, 4, 7 and 10) and washout week (3, 6 and 9)
  Severity of fatigue will be evaluated by the Daily-Fatigue Impact Scale (D-FIS), a questionnaire containing 8 items that evaluates the impact of fatigue on cognition, physical functioning, and daily activities.

OTHER OUTCOMES:
Measurement of biomarkers as in detailed description of the study section | These will be measured singularly during baseline week (0)
  Measurement of specific biomarkers will be performed in order to enable us to characterise individuals with self-reported non-coeliac gluten sensitivity

CONTACTS AND LOCATIONS:
Locations (1):
- University of Aberdeen Rowett Institute of Nutrition and Health, Aberdeen, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Rees D, Holtrop G, Chope G, Moar KM, Cruickshank M, Hoggard N. A randomised, double-blind, cross-over trial to evaluate bread, in which gluten has been pre-digested by prolyl endoprotease treatment, in subjects self-reporting benefits of adopting a gluten-free or low-gluten diet. Br J Nutr. 2018 Mar;119(5):496-506. doi: 10.1017/S0007114517003749. PMID 29508689